CLINICAL TRIAL: NCT00925132
Title: Phase Ib/II: Epigenetic Modification of Chemosensitivity and Apoptosis in Metastatic Melanoma: Treatment of a Resistant Disease Using Decitabine, Temozolomide and Panobinostat
Brief Title: Treatment of Resistant Metastatic Melanoma Using Decitabine, Temozolomide and Panobinostat
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in the number of approved drugs for metastatic melanoma
Sponsor: University of Iowa (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mohammed M Milhem, Clinical Associate Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200807728
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic; Melanoma; Epigenetic; Temozolomide; Decitabine; Panobinostat; LBH589
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Temozolomide; Decitabine; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide, Decitabine, Panobinostat (Experimental): Temozolomide - given each cycle.
  Decitabine - 6 cohorts with dose escalation.
  Panobinostat - 6 cohorts with dose escalation.
  Interventions: Drug: Temozolomide, Decitabine, Panobinostat

INTERVENTIONS:
Drug: Temozolomide, Decitabine, Panobinostat — Temozolomide - given each cycle.
  Decitabine - 6 cohorts with dose escalation.
  Panobinostat - 6 cohorts with dose escalation.
  Other Names: LBH589

SUMMARY:
The purpose of this study is to treat metastatic melanoma with a combination of standard chemotherapy (decitabine and Temozolomide in a dose escalation scheme) with an study drug called panobinostat. This combination is proposed to unlock genes that may contribute to mechanisms that cause tumor growth.

The primary objectives of this study are:

* To evaluate the safety and tolerability of the proposed schedule of decitabine, temozolomide and panobinostat in the treatment of metastatic melanoma.
* To define any Dose Limiting Toxicity (DLT) and maximum tolerated dose (MTD) of the combination of decitabine, temozolomide and panobinostat.

DETAILED DESCRIPTION:
Most chemotherapeutics target rapidly proliferating cells, leaving quiescent cells and those with extended cell cycles unaffected. The investigators propose that this combination of decitabine, temozolomide, and panobinostat will target both melanoma stem cells and rapidly proliferating melanoma cells. The use of two drugs that regulate gene expression epigenetically (panobinostat and decitabine) in combination with a chemotherapeutic agent (temozolomide) is hypothesized to:

* induce expression genes (e.g., Apaf-1) that increase chemosensitivity of tumor cells and enhance apoptosis
* potentiate the cytotoxic effect of temozolomide by epigenetic modulation, and
* induce proliferation and differentiation of tumor stem cells, thus enabling senescence and apoptosis.

Secondary objectives:

* To measure overall survival
* To measure the time to progression of patients treated with this combination in comparison to patients treated historically with DTIC (the current standard of care).
* To evaluate treatment response with FDG PET and compare FDG PET with conventional imaging for treatment response assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old
2. ECOG Performance Status of ≤ 2
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
4. Patients must have measurable disease according to RECIST and CHOI criteria. The minimum target-lesion diameter should have double the CT slice thickness, i.e., 10 mm
5. Patients must meet the following laboratory criteria:

   Hematology: Neutrophil count of >1500/mm3;Platelet count of > 100,000/mm3L; Hemoglobin ≥ 9 g/dL Biochemistry:AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x upper limit of normal if the transaminase elevation is due to disease involvement;Serum bilirubin ≤ 1.5 x upper limit of normal;Serum creatinine ≤ 1.5 x upper limit of normal or 24-hour creatinine clearance ≥ 50 ml/min; Total serum calcium (corrected for serum albumin) or ionized calcium ≥ lower limit of normal; Serum potassium ≥ lower limit of normal; Serum sodium ≥ lower limit of normal;Serum albumin ≥ lower limit of normal or 3g/dl;Patients with any elevated alkaline phosphatase due to bone metastasis can be enrolled
6. Baseline ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal.
7. TSH and free T4 within normal limits (patients may be on thyroid hormone replacement)
8. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 8 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
9. Any patient with the diagnosis of metastatic melanoma from any site. These include untreated patients or those treated with chemotherapy or biochemotherapy.
10. Must not have taken a hypomethylating agent or a histone deacetylase agent in the treatment of their disease. Patients who receive targeted agents would only need a 2-week washout period.
11. Any patient with metastatic melanoma regardless of prior treatment will be eligible.
12. Patients must have had disease progression on or following their most recent treatment regimen or on presentation for the first time with metastatic disease, surgical option can be entertained if this is a localized relapse.
13. Patients with CNS disease are eligible for treatment only after their CNS disease has been directly addressed with radiation therapy.

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
2. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
3. Impaired cardiac function including any one of the following: Screening ECG with a QTc > 450 msec confirmed by central laboratory prior to enrollment to the study; Patients with congenital long QT syndrome; History of sustained ventricular tachycardia; Any history of ventricular fibrillation or torsades de pointes; Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible; Patients with a myocardial infarction or unstable angina within 6 months of study entry; Congestive heart failure (NY Heart Association class III or IV);Right bundle branch block and left anterior hemiblock (bifascicular block)
4. Uncontrolled hypertension
5. Concomitant use of drugs with a risk of causing torsades de pointes
6. Concomitant use of CYP3A4 inhibitors
7. Patients with unresolved diarrhea > CTCAE grade 1
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat
9. Other concurrent severe and/or uncontrolled medical conditions
10. Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
11. Concomitant use of any anti-cancer therapy or radiation therapy.
12. Patients who have no measurable disease.
13. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP)not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months(i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 8 days of the first administration of oral panobinostat.
14. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
15. Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
16. Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
17. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia C, Leon-Ferre R, Laux D, Deutsch J, Smith BJ, Frees M, Milhem M. Treatment of resistant metastatic melanoma using sequential epigenetic therapy (decitabine and panobinostat) combined with chemotherapy (temozolomide). Cancer Chemother Pharmacol. 2014 Oct;74(4):691-7. doi: 10.1007/s00280-014-2501-1. Epub 2014 Jul 26. PMID 25062770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between December 2009 through June 2015. The study population was accessed via the Principal Investigator's medical clinic at Holden Comprehensive Cancer Center.
Pre-assignment Details: Following consent, all subjects undergo screening procedures to verify eligibility for participation in the study. Screening included physical exam, blood and urine tests to check general health, blood test for fetal hemoglobin, blood test for pregnancy (only for women of childbearing age), ECG and Echo, CT and FDG-PET, and tumor measurements
Groups:
- Phase I:Decitabine 0.1mg/kg + Panobinostat 10mg + Temozolomide: Cohort 1: Participants were administered Decitabine 0.1 mg/kg via subcutaneous injection (SQ) 3x weekly, Panobinostat 10mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
- Phase I:Decitabine 0.1 mg/kg + Panobinostat 20mg +Temozolomide: Cohort 2: Participants were administered Decitabine 0.1 mg/kg via subcutaneous injection (SQ) 3x weekly, Panobinostat 20mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
- Phase I:Decitabine 0.2 mg/kg + Panobinostat 20mg+Temozolomide: Cohort 3: Participants were administered Decitabine 0.2 mg/kg via subcutaneous injection (SQ) 3x weekly, Panobinostat 20mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
- Phase I:Decitabine 0.2 mg/kg + Panobinostat 30mg +Temozolomide: Cohort 4: Participants were administered Decitabine 0.2 mg/kg via subcutaneous injection (SQ) 3x weekly and Panobinostat 30mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
- Phase II:Decitabine 0.2 mg/kg+Panobinostat 30mg+Temozolomide: Participants were administered Decitabine 0.2 mg/kg via subcutaneous injection (SQ) 3x weekly and Panobinostat 30mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
Period: Overall Study
Arm/Group | Phase I:Decitabine 0.1mg/kg + Panobinostat 10mg + Temozolomide | Phase I:Decitabine 0.1 mg/kg + Panobinostat 20mg +Temozolomide | Phase I:Decitabine 0.2 mg/kg + Panobinostat 20mg+Temozolomide | Phase I:Decitabine 0.2 mg/kg + Panobinostat 30mg +Temozolomide | Phase II:Decitabine 0.2 mg/kg+Panobinostat 30mg+Temozolomide
Started | 5 | 4 | 4 | 4 | 22
Completed | 3 | 4 | 4 | 4 | 17
Not Completed | 2 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1
Not completed — Removed due to disease progression | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Patients with the diagnosis of metastatic melanoma from any site. These include untreated patients or those treated with chemotherapy or biochemotherapy.
Groups:
- Temozolomide, Decitabine, Panobinostat: Temozolomide - given each cycle.
  Decitabine - 6 cohorts with dose escalation.
  Panobinostat - 6 cohorts with dose escalation.
  Temozolomide, Decitabine, Panobinostat: Temozolomide - given each cycle.
  Decitabine - 6 cohorts with dose escalation.
  Panobinostat - 6 cohorts with dose escalation.
Arm/Group | Temozolomide, Decitabine, Panobinostat
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 37
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Number of Participants With Dose Limiting Toxicities (DLTs) at a Given Dose Level
Description: A DLT was any Grade 4 toxicity for neutrophils or platelets for ≥ 7 days, Grade 3 toxicity for neutrophils for ≥ 21 days, any Grade 3 solid organ toxicity not explainable by another cause (e.g. neurotoxicity, GI toxicity), metabolic/laboratory toxicity (≥10 x ULN AST) for ≥ 14 days, any Grade 4 infection or QTcF> 500msec EKG. DLTs were assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0.
  All adverse events were collected and graded to determine DLTs as assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0. DLTs were assessed to determine the recommended Decitabine and Panobinostat dose for the Phase II portion of the trial.
Time Frame: 6 weeks (one full cycle)
Population: Number of patients within the 4 dosing cohorts evaluable for DLTs following administration of one full cycle
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Escalation: Temozolomide - given each cycle.
  Decitabine - 6 cohorts with dose escalation.
  Panobinostat - 6 cohorts with dose escalation.
Arm/Group | Phase I Dose Escalation
Number analyzed (Participants) | 15
Participants
  Cohort 1: Experienced DLT | 0
  Cohort 2: Experienced DLT | 0
  Cohort 3: Experienced DLT | 0
  Cohort 4: Experienced DLT | 0

2. Primary Outcome: Phase 2 -Number of Patients With a Decrease in Tumor Size Using RECIST and CHOI's Criteria
Description: Tumor response rate was assessed using RECIST criteria in which a complete response was the disappearance of all target lesions; Partial response was a 30% decrease in the sum of the longest dimension (LD) of target lesions, relative to baseline measurement; Progressive disease was an increase of 20% or more in the sum of the LD of target lesions; and Stable disease was a decrease in tumor size of less than 30% or increase of less than 20%.
  Tumor response rate was also assessed using CHOI's criteria in which a response was a 10% decrease in tumor size or a 15% decrease in tumor density on contrast-enhanced computed tomography scan.
  Tumor response rates were assessed in order to determine effectiveness of the treatment regimen which was defined by the response rate of at least 30% as measured by either the RECIST or Choi's criteria, and ineffective if the rate is less than 15% on both.
Time Frame: 12 weeks (2 cycles)
Population: Number of patients evaluable for tumor response assessment following 2 cycles of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Phase II:Decitabine 0.2 mg/kg +Panobinostat 30mg +Temozolomide: Participants were administered Decitabine 0.2 mg/kg via subcutaneous injection (SQ) 3x weekly, Panobinostat 30mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
Arm/Group | Phase II:Decitabine 0.2 mg/kg +Panobinostat 30mg +Temozolomide
Number analyzed (Participants) | 17
Participants
  Progressive Disease (PD) | 12
  Stable Disease (SD) | 5

3. Secondary Outcome: Phase 2 - Number of Participants With Disease Progression
Description: Number of participants who died or had disease progression
Time Frame: 5 years
Population: Number patients who received study drug in Phase II portion of trial
Measure: Count of Participants; unit: Participants
Groups:
- Phase II:Decitabine 0.2 mg/kg +Panobinostat 30mg+Temozolomide: Participants were administered Decitabine 0.2 mg/kg via subcutaneous injection (SQ) 3x weekly and Panobinostat 30mg orally (PO) once every 96 hours for 2 weeks and Temozolomide at a dose of 150 mg/m2 orally Day 9 through 13 for 5 doses. Dose for Temozolomide was escalated to 200 mg/m2 for 5 days after Cycle 1.
Arm/Group | Phase II:Decitabine 0.2 mg/kg +Panobinostat 30mg+Temozolomide
Number analyzed (Participants) | 22
Participants
  Died within 5 year time frame | 17
  Removed due to disease progression | 5

ADVERSE EVENTS:
Arm/Group | Temozolomide, Decitabine, Panobinostat
Serious Adverse Events (participants affected / at risk) | 5/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide, Decitabine, Panobinostat (N=39)
Obstruction, GI (small bowel) (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Obstruction, GU (ureter) (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema-lower extremity (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide, Decitabine, Panobinostat (N=39)
Leukocytes (Blood and lymphatic system disorders) | 24 (24)
Lymphopenia (Blood and lymphatic system disorders) | 29 (29)
RBC Decreased (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 14 (14)
Neutrophils (Blood and lymphatic system disorders) | 27 (27)
Platelets (Blood and lymphatic system disorders) | 24 (24)
Fatigue (General disorders) | 24 (24)
Fever (General disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 22 (22)
Vomiting (Gastrointestinal disorders) | 11 (11)
Tachycardia (Cardiac disorders) | 3 (3)
ALT (Metabolism and nutrition disorders) | 11 (11)
Albumin (Metabolism and nutrition disorders) | 1 (1)
Bicarbonate-Serum low (Metabolism and nutrition disorders) | 4 (4)
Bilirubin (Metabolism and nutrition disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 3 (3)
GGT (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (14)
Chloride decreased (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 6 (6)
Left Sided Weakness (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 8 (8)
Hyponatremia (Metabolism and nutrition disorders) | 10 (10)
Headache (General disorders) | 3 (3)
Anxiety (Nervous system disorders) | 2 (2)
Coagulation PTT (Blood and lymphatic system disorders) | 1 (1)
Failure to thrive (General disorders) | 1 (1)
Albumin-Serum low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (7)
Potassium-Serum low (hypokalemia) (Metabolism and nutrition disorders) | 6 (6)
Phosphorous (Metabolism and nutrition disorders) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (General disorders) | 2 (2)
Neuropathy (General disorders) | 2 (2)
Weight Loss (Metabolism and nutrition disorders) | 3 (3)
Insomnia (General disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Speech impairment (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
General pain: chest and body (Musculoskeletal and connective tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Gastritis (Gastrointestinal disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 (6)
Somnolence (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was closed to enrollment early as there was a change in the number of approved drugs for metastatic melanoma, making Temozolomide as a chemotherapy agent, an unlikely treatment for metastatic melanoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes